CLINICAL TRIAL: NCT02282969
Title: Promoting Informed Decisions About Lung Cancer Screening: Decision Aid Update and Measures Development
Brief Title: PCORI-CER-1306-03385 Lung Cancer Screening Decision Aid Development and Testing
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PA14-0072; CER-1306-03385 (Other Grant/Funding Number: Patient Centered Outcomes Research Institute); NCI-2022-00832 (Other: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2014-10-31; First posted 2014-11-05 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Health Knowledge, Attitudes, Practice
Keywords: Cancer Prevention; Smokers; Quit smoking; Interviews; Questionnaires; Surveys; Lung cancer screening; Patient decision aid
MeSH Terms: conditions — Behavior | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung Cancer Screening Decision Aids: Participants are asked to look over education materials about lung cancer screening, and interviewed. Some participants will look at a video patient decision aid, with an interview and questionnaire completion. Some participants complete lung cancer screening knowledge questionnaire at first visit, and then again in one month.
  Interventions: Behavioral: Interviews; Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Interviews — Interviews performed by study staff encompassing lung cancer screening and patient decision aids.
Behavioral: Questionnaires — Questionnaires completed after viewing patient decision aid video. Questionnaires also completed regarding lung cancer screening knowledge at first visit, then again in one month.
  Other Names: Surveys

SUMMARY:
Objectives:

This protocol addresses the first phase of a larger project funded by the Patient-Centered Outcomes Research Institute to help heavy smokers make informed decisions about lung cancer screening with low-dose computed tomography (CT). A separate IRB protocol will be submitted for the larger, comparative study. In this initial development phase, our prototype patient decision aid will be updated to reflect current guidelines about lung cancer screening. The updated aid will then be pilot-tested in a new sample of patients. In addition, several of the study measures will be refined and further developed in preparation for the larger study.

The specific aims of the measures and decision aid development phase of this project are as follows:

Update the aid to reflect current screening guidelines and refine the aid via cognitive testing with patients/smokers; and pilot test the updated aid for acceptability with patients/smokers.

Modify our current measure of lung cancer knowledge, conduct cognitive testing of the new measure with patients/smokers, and evaluate the reliability of the new measure in a sample patients/smokers.

DETAILED DESCRIPTION:
Cognitive and Pilot Testing:

If you agree to take part in this study, you will take part in an interview with a member of the research staff. The interviewer will take notes of your responses. First, you will be asked some questions about you, like your age, sex, race, and education level. Then you will be asked to look at some educational materials about lung cancer screening. These could be written information, animations, graphics, videos, or questionnaires. You may be asked questions about:

* Lung cancer and lung cancer screening
* The length of the materials
* The balance of the information found in the materials

The study interview will take place in person at MD Anderson and will take between 1 and 1 ½ hours.

Your participation on this study will be over once the interview is complete.

This is an investigational study.

Up to 50 participants will be enrolled in this part of the study. All will take part at MD Anderson, UTMB, the Galveston community, or tobacco-related community events.

Measures Reliability Study:

If you agree to take part in this study, you will complete a questionnaire 2 times. The questionnaire will ask about:

* Lung cancer
* Lung cancer screening
* Making decisions about screening
* Your age, race, gender, and level of education

You will complete the first questionnaire in person. It will take about 20 minutes to fill out. Then, about 1 month later, you will be asked to fill out the questionnaire again.

The second time you can come in person, or fill out the questionnaire by mail or telephone. Your participation will be over when the second questionnaire is complete.

This is an investigational study.

Up to 150 participants will be enrolled in this part of the study. All will take part at MD Anderson, UTMB, the Galveston community, or tobacco-related community events.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 55 to 80 years of age.
2. Participants must speak English.
3. Current smoker or quit smoking within the past 15 years.

Exclusion Criteria:

1. History of lung cancer.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants recruited from Houston and Galveston areas.
Sampling Method: Non-Probability Sample
Enrollment: 620 (Estimated)
Dates: Start 2014-07-11 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Informed Decisions About Lung Cancer Screening (Data from interviews and questionnaires reviewed to assess participant knowledge) | 1 Month
  Data from interviews and questionnaires reviewed to assess participant knowledge regarding lung cancer screening and decision aid.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Volk, PHD, Study Chair — M.D. Anderson Cancer Center; Suzanne Linder, PHD, Principal Investigator — The University of Texas Medical Branch at Galveston; Paul Cinciripini, PHD, MS, BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - The University of Texas Medical Branch at Galveston, Galveston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org